CLINICAL TRIAL: NCT04154891
Title: Etude Pilote Des différentes stratégies de séquençage Haut débit du génome Pour le Diagnostic génétique Des Patients Atteints de déficience Intellectuelle
Brief Title: Genome Sequencing Strategies for Genetics Diagnosis of Patients With Intellectual Disability
Acronym: DEFIDIAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Commissariat A L'energie Atomique (Other Government); Hospices Civils de Lyon (Other); Centre Hospitalier Universitaire Dijon (Other); University Hospital, Rouen (Other); University Hospital, Strasbourg (Other); APHP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: C16-110; 2018-A00680-55 (Other: IDRCB)
Record Dates: First submitted 2019-10-29; First posted 2019-11-07 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Intellectual Disability
Keywords: Rare disease; Next generation sequencing genome; Diagnostic study; Medico-economic study
MeSH Terms: conditions — Intellectual Disability; Rare Diseases; Disease

STUDY DESIGN:
Intervention Model Description: Prospective multicenter diagnostic study comparing the percentage of Intellectual Deficiency (ID) causal diagnosis obtained using 2 main different strategies (Whole Genome Sequencing using a trio strategy (WGST), and reference strategy) applied blindly to consecutive patients with no obvious diagnosis. Each included patient will be his own control; he will benefit from the two main strategies compared, in parallel. The diagnostic yield of Whole Genome Sequencing using a simplex strategy (WGSs) will be also investigated in parallel to the two main strategies but only in a randomized subgroup of the overall population coming for a first genetic advice.
Who Masked: Outcomes Assessor
Masking Description: The results of the different strategies will be interpreted blindly, each participating laboratory being in charge for a given investigation center, either of 1) the trio or 2) the 44GPS (part of the reference strategy) and, for the randomized sub-population of the overall population coming for a first genetic advice, simplex analyses. Fra-X and chromosomal microarray analysis corresponding to the reference strategy will follow the routine circuit, which is mainly independent from the WGS circuit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Trio Whole Genome Sequencing — WGS trio analysis will be performed using the genome data of the index case in addition to the genome data of his parents. This analysis will follow a consensus protocol that contains 3 obligatory steps: first of all, de novo variants (SNV, CNV and others SV) will be examined in the whole genome data set; then, a SNV/CNV/other SV analysis will be performed under a AR or X linked Mendelian mode hypothesis in the whole genomic regions of a OMIM extended list (that contains all genes already involved in human genetic diseases). Finally, analysis will focus on inherited pathogenic variants under an AD mode hypothesis (analysis of variations already reported as pathogenic in clinVar or HGMD pro; CNV or truncating variation in OMIM genes, etc). When these 3 steps analysis is completed then variants of interest identified at each step will be recorded until examination by a specific multidisciplinary meeting.
Genetic: Simplex Whole Genome Sequencing — This analysis will be performed using only the index case following a similar strategy than the one used for the WGS trio
Genetic: Current French Reference strategy — Actual ANPGM recommendations defined by the following analysis: Fra-X + chromosomal microarray analysis + 44GPS

SUMMARY:
Introduction : Intellectual Disability (ID) is the most common cause of referral in the pediatric genetic centers and is characterized by an extreme genetic heterogeneity corresponding to a myriad of rare diseases that complicates the identification of ID's.

Overall today in France, for non-syndromic ID affected patients, the Fra-X detection, the chromosomal microarray analysis and Gene Panel Strategy of 44 ID selected genes leads to a global diagnostic yield for 1/3 patients leaving 2/3 of patients still with no diagnosis.

The advent, and burst, of Next Generation Sequencing (NGS) technologies has clearly revolutionized the approaches to diagnosis and research in the field of rare diseases at an international. That's why the main hypothesis of DEFIDIAG is that Whole Genome Sequencing (WGS) could allow to improve the diagnostic performance and cost-effectiveness for French patients with ID.

Objective : The main objective of this study is to compare ther percentage of genetic causal diagnosis identified in ID patients by performing trio WGS analysis vs the use of the current French reference strategy (ACPA, X-Fra, DI 44).

Methods and design : This is a prospective study. The investigators expect to include 1275 index case with his/her 2 biological unaffected parents.

ELIGIBILITY:
1. Inclusion criteria for children or adults with ID of unknown etiology (index case)

   In order to be eligible to participate in this study, an individual must meet all the following criteria:
   * Age:

     1. Between 0 and 5 years with stringent criteria (severe delayed development in terms of motor skills, language, and/or sociability) OR
     2. ≥ 6 years: patients with ID, whatever the severity (but with proven ID by ad hoc neuropsychological testing) and the associated manifestations
   * Without any obvious diagnosis identified during a genetic consultation in one of the participating center (i.e., an obvious syndrome with ID with well-known molecular diagnosis is excluded);
   * Provision of signed and dated of "participant" consent form;
   * Stated willingness to comply with all study procedures and availability for the duration of the study.

   Patient with a social security in compliance with the French law (Provisions relating to research involving the human person provided for in Articles L 1121-1 et seq. of the French Public Health Code).
2. Inclusion criteria for biological parents

   - Provision of signed and dated of both parents consent form.
3. Non-inclusion criteria

   * An individual, who presents any condition which in the investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol, will not be eligible;
   * Patients with isolated learning disabilities;
   * One or both parents with ID;
   * Parent placed under judicial protection (tutelle, curatelle et sauvegarde de justice) ;
   * Patient with a known etiological diagnosis (non-genetic, previously proven Fra-X syndrome, know chromosomal anomaly, known pathogenic or probably pathogenic variant identified in an ID gene by any technique).
   * For patient concerning by biobank project: hypersensitivity to local anesthesia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3825 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Diagnostic Yield | 12 months
  The primary study endpoint is the identification of a causal diagnosis of ID defined as the identification of one class 4 or 5 variant (or two in case of autosomal recessive inheritance) that explains the symptoms presented by the patient. In addition variants classified as 3+, anticipated to become future 4 will be recorded. Specific analysis and follow up of the variant classified as 3+ (i.e. with a high probability of pathogenicity) will be done after the end of the protocol to determine the class 3+ to class 4-5 switch proportion and to describe the new genes/mechanisms involved in ID and revealed by DEFIDIAG.

SECONDARY OUTCOMES:
Causal structural change | 12 months
  Identification of causal structural changes (CNV, translocation, inversion) in the first investigation population (confirmed during the MDM for the WGS strategies)
  The clinical characteristics of patients and the diagnostic yield at each step of the incremental selection within WGS analyses (44GPS, OMIMOME, WES, WGS) according to the results of the preceding step as well as according to the results of chromosomal microarray analysis and 44GPS will also be parameters of interest in the whole population.
Incremental cost-effectiveness ratio | 24 months
  The cost-effectiveness endpoint will be an efficiency criterion based on the estimation of an incremental cost-effectiveness ratio, expressed in terms of cost per additional positive diagnosis.
Mean cost of wavering diagnostic research | 24 months
  Estimation of the cost of wavering diagnostic research
Percentage of at least one modification in medical, medico-social, rehabilitative and psychological follow-up | 24 months
Number and type of secondary data | 12 months
  The number and type of SFs (class 4 or 5 mutation(s)) identified in the parents that specifically consent to this study will be recorded in a specific report. The outcome will be defined by the percentage of SFs in the studied population and the number and type of medical consequences following their identification.
Median time and type of skills required for analyzing genetic data and for genetic confirmation | 12 months
Median time to obtain results | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hélène DOLLFUS, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (14):
- France (14):
  - CHU d'Angers, Angers
  - CHU Bordeaux, Bordeaux
  - Hospices Civil de Lyon, Bron
  - CHU Dijon, Dijon
  - CHU de Grenoble-Alpes, La Tronche
  - CHRU Lille, Lille
  - Assistance publique - Hôpitaux de Marseille, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Assistance publique - Hôpitaux de Paris - Groupe Hospitalier Pitié Salpétrière, Paris
  - Assistance publique - Hôpitaux de Paris - Hôpital Necker - Enfants malades, Paris
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU Strasbourg, Strasbourg

REFERENCES:
- [Background] Binquet C, Lejeune C, Faivre L, Bouctot M, Asensio ML, Simon A, Deleuze JF, Boland A, Guillemin F, Seror V, Delmas C, Esperou H, Duffourd Y, Lyonnet S, Odent S, Heron D, Sanlaville D, Frebourg T, Gerard B, Dollfus H. Genome Sequencing for Genetics Diagnosis of Patients With Intellectual Disability: The DEFIDIAG Study. Front Genet. 2022 Feb 1;12:766964. doi: 10.3389/fgene.2021.766964. eCollection 2021. PMID 35178068
- [Background] Lejeune C, Robert-Viard C, Meunier-Beillard N, Borel MA, Gourves L, Staraci S, Soilly AL, Guillemin F, Seror V, Achit H, Bouctot M, Asensio ML, Briffaut AS, Delmas C, Bruel AL, Benoit A, Simon A, Gerard B, Hadj Abdallah H, Lyonnet S, Faivre L, Thauvin-Robinet C, Odent S, Heron D, Sanlaville D, Frebourg T, Muller J, Duffourd Y, Boland A, Deleuze JF, Esperou H, Binquet C, Dollfus H. The Economic, Medical and Psychosocial Consequences of Whole Genome Sequencing for the Genetic Diagnosis of Patients With Intellectual Disability: The DEFIDIAG Study Protocol. Front Genet. 2022 Apr 4;13:852472. doi: 10.3389/fgene.2022.852472. eCollection 2022. PMID 35444683
- [Background] Meuwissen M, Verstraeten A, Ranza E, Iwaszkiewicz J, Bastiaansen M, Mateiu L, Nemegeer M, Meester JAN, Afenjar A, Amaral M, Ballhausen D, Barnett S, Barth M, Asselbergh B, Spaas K, Heeman B, Bassetti J, Blackburn P, Schaer M, Blanc X, Zoete V, Casas K, Courtin T, Doummar D, Guerry F, Keren B, Pappas J, Rabin R, Begtrup A, Shinawi M, Vulto-van Silfhout AT, Kleefstra T, Wagner M, Ziegler A, Schaefer E, Gerard B, De Bie CI, Holwerda SJB, Abbot MA, Antonarakis SE, Loeys B. Heterozygous variants in CTR9, which encodes a major component of the PAF1 complex, are associated with a neurodevelopmental disorder. Genet Med. 2022 Jul;24(7):1583-1591. doi: 10.1016/j.gim.2022.04.003. Epub 2022 May 2. PMID 35499524
- [Background] Ravindran E, Lesca G, Januel L, Goldgruber L, Dickmanns A, Margot H, Kaindl AM. Case report: Compound heterozygous NUP85 variants cause autosomal recessive primary microcephaly. Front Neurol. 2023 Feb 9;14:1124886. doi: 10.3389/fneur.2023.1124886. eCollection 2023. PMID 36846113
- [Derived] El Chehadeh S, Heide S, Quelin C, Rio M, Margot H, Genevieve D, Isidor B, Goldenberg A, Guegan C, Lesca G, Willems M, Ormieres C, Caumes R, Busa T, Bonneau D, Guerrot AM, Marey I, Vera G, Marzin P, Philippe A, Garde A, Coubes C, Vincent M, Michaud V, Mignot C, Charles P, Sigaudy S, Edery P, Lacombe D, Boland A, Nowak F, Bouctot M, Humbert-Asensio ML, Simon A, Chennen K, Sabour N, Delmas C, Nicolas G, Saugier-Veber P, Lecoquierre F, Cassinari K, Keren B, Courtin T, De Sainte Agathe JM, Malan V, Barcia G, Tran Mau-Them F, Safraou H, Philippe C, Thevenon J, Chatron N, Januel L, Piton A, Haushalter V, Gerard B, Lejeune C, Faivre L, Sanlaville D, Heron D, Odent S, Nitschke P, Schluth-Bolard C, Lyonnet S, Deleuze JF, Binquet C, Dollfus H; DEFIDIAG study group. Genome sequencing for the diagnosis of intellectual disability as a paradigm for rare diseases in the French healthcare setting: the prospective DEFIDIAG study. Genome Med. 2025 Oct 3;17(1):110. doi: 10.1186/s13073-025-01527-4. PMID 41044778